CLINICAL TRIAL: NCT03026751
Title: Improving Diagnosis in Idiopathic Cytopenia Using Gene Sequencing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4384
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Next-generation sequencing will occur looking at target genes in the marrow to identify mutations.
  DNA will be sequenced to allow us to determine acquired mutations in haematopoietic tissue.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bone Marrow Aspirate — Bone marrow aspirate

SUMMARY:
10% of the cases referred to the specialist diagnostic haemato-pathology service at RMH are for cytopenias.

The hypothesis to be tested is that a proportion of patients with idiopathic cytopenias have mutations in myelodysplasic syndrome (MDS)-associated genes. The investigators will sequence a panel of known MDS-associated genes in patient material (bone marrow and blood) that is sent routinely to the diagnostic service where conventional techniques have failed to establish a clear diagnosis. 200 patients with idiopathic cytopenia will be followed up to determine their survival, blood counts and development of acute leukaemia and other haematological malignancies. The clinical outcomes will be correlated with any mutations detected.

DETAILED DESCRIPTION:
Patients with cytopenias will be identified by their local District General Consultant haematologist and consent obtained. A bone marrow sample will be sent to RMH as per usual diagnostic pathway.

Once received at the RMH, an aliquot will be frozen down for sequencing by the Molecular Pathology lab. Only those cases of cytopenia without a specific diagnosis will be the focus of this study.

Results will be fed back to referring consultants with caveats regarding significance.

Patients will undergo telephone follow up and data will also be provided by local consultants.

The investigators will look at overall survival, development of haematological malignancies and full blood count. This will occur annually.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients >= 18 years old
* Life expectancy more than 12 months
* Cytopenia defined as Hb < 110g/L and/or Neutrophils <1.5 x109/L and/or Platelets <100 x109/L

Exclusion Criteria:

* Known haematological malignancy or aplastic anaemia/paroxysmal nocturnal haemoglobinuria
* Cytopenia of known aetiology (after examination of blood film and other investigations have occurred). These include haematinic deficiency (patients unresponsive to appropriate haematinic deficiency may enter the study), autoimmune cytopenias, chronic renal anaemia (for those with isolated anaemia), known haemoglobinopathy (for those with isolated anaemia), chronic viral diseases (Hep B/C/HIV), cytopenias associated with liver disease, cytopenias associated with systemic autoimmune conditions (eg SLE, rheumatoid arthritis), anaemia of chronic disease (for those with isolated anaemia).
* Cytotoxic chemotherapy or other myelosuppressive drugs or radiotherapy within 12 months
* Inadequate bone marrow sample for gene testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood and bone marrow samples are routinely sent to RMH from District General Hospitals for special tests to make a diagnosis for patients with blood problems.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with idiopathic cytopenia with a mutation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Taussig, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No